CLINICAL TRIAL: NCT05083026
Title: Neutralizing Antibody Level After COVID-19 Vaccination in Hospital Works.
Brief Title: Neutralizing Antibody Level After COVID-19 Vaccination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Su Youn Nam, Assistant professor, Kyungpook National University Hospital
Other Study IDs: KNUCH-2021005-001-001
Record Dates: First submitted 2021-08-08; First posted 2021-10-19 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. 5mL blood at 2, 4, 6, 9, 12 months after COVID-19 vaccination.
  2. centrifuge and get serum sample
  3. store at -80 degree deep freezer until use
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COVID-19 neutralizing antibody — This study enrolled persons already who received COVID-19 vaccination under government policy.
  1. We collect 5mL blood at 2, 4, 6, 9, 12 months after COVID-19 vaccination
  2. isolate serum and store in -80 degree deep freezer
  3. measure neutralizing Antibody

SUMMARY:
1. serial of neutralizing antibody at 2, 4, 6, 9, 12 month after COVID-19 vaccination
2. investigate the factors on antibody titer.

DETAILED DESCRIPTION:
1. serial of neutralizing antibody at 2, 4, 6, 9, 12 month after COVID-19 vaccination 1) semi-quantitative measurement of neutralizing antibody at 2, 4, 6, 9, 12 month after COVID-19 vaccination 2) investigate the duration maintaining acceptable range (over 30% inhibition)
2. investigate the factors on antibody titer at 2 month after vaccination 1) potential factors: age, sex, body weight, height, use of medication, use of antipyretics (NSAID or tyrenol), side effect of COVID-19 vaccination 2) correlation between antibody titer and potential factors
3. Compare 4 diagnostic ELISA kit at 2 month after vaccination 1) measure neutralizung antibody using ELISA kits from 4 different companies 2) investigate correlation coefficient of antibody titer between companies

ELIGIBILITY:
Inclusion Criteria:

* healthcare works after completion of COVID-19 vaccination
* 20-60 years
* sign the agreement of study

Exclusion Criteria:

* serious underlying diseases

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: healthcare works aged 20-60 years after completion of COVID-19 vaccination
  participants have no serious disease.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
titer of neutralizing antibody after COVID-19 vaccination | at 2month after COVID-19 vaccination
  semi-quantitative measurement of neutralizing antibody after COVID-19 vaccination
titer of neutralizing antibody after COVID-19 vaccination | at 4 month after COVID-19 vaccination
  semi-quantitative measurement of neutralizing antibody after COVID-19 vaccination
titer of neutralizing antibody after COVID-19 vaccination | at 6 month after COVID-19 vaccination
  semi-quantitative measurement of neutralizing antibody after COVID-19 vaccination
titer of neutralizing antibody after COVID-19 vaccination | at 9 month after COVID-19 vaccination
  semi-quantitative measurement of neutralizing antibody after COVID-19 vaccination
titer of neutralizing antibody after COVID-19 vaccination | at 12 month after COVID-19 vaccination
  semi-quantitative measurement of neutralizing antibody after COVID-19 vaccination
body weight (Kg) | at 2 month after COVID-19 vaccination
  correlation between antibody titer and body weight: spearmann's correlation
body mass index (kg/m^2) | at 2 month after COVID-19 vaccination
  correlation between antibody titer and body weight: spearmann's correlation
Compare 4 diagnostic ELISA kit after COVID-19 vaccination | at 2 month after COVID-19 vaccination
  1. measure neutralizung antibody using ELISA kits from 4 different companies 2 months after COVID-19 vaccination
  2. investigate correlation coefficient of antibody titer between companies

CONTACTS AND LOCATIONS:
Overall Officials: Su Youn Nam, MD, PhD, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nam SY, Jeon SW, Jung DK, Heo SJ. Body Weight is Inversely Associated with Anti-SARS-CoV-2 Antibody Levels after BNT162b2 mRNA Vaccination in Young and Middle Aged Adults. Infect Chemother. 2022 Sep;54(3):504-516. doi: 10.3947/ic.2022.0089. PMID 36196609